CLINICAL TRIAL: NCT01383681
Title: Observational Study To Establish The Methodology Used In The Evaluation, Treatment And Assessment Of Progression Of Spasticity In The Spanish Population
Brief Title: Retrospective Study of Patients With Spasticity in the Spanish Population
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/NS/SPA/019
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-09

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: This was a retrospective chart review in patients with spasticity in the Spanish population. There was no treatment in this study.
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — There was no treatment in this study.

SUMMARY:
This is a retrospective study of patients with spasticity in the Spanish population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spasticity

Exclusion Criteria:

* Current enrollment in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of spasticity are selected from rehabilitation departments within the Spanish health system.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Mataró, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a retrospective chart review in patients with spasticity in the Spanish population.
Period: Overall Study
Arm/Group | All Participants
Started | 235
Completed | 189
Not Completed | 46

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 235
Age, Customized [Number; unit: Participants]
  18 to 25 years | 21
  26 to 35 years | 21
  36 to 45 years | 43
  46 to 55 years | 48
  56 to 65 years | 57
  >65 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 141

OUTCOME MEASURES:

1. Primary Outcome: Physician Assessment of Spasticity
Description: The physician assessed spasticity as per local standard practice. Not enough data was collected for analysis of this outcome measure.
Time Frame: Baseline
Population: Planned analysis: All participants. Not enough data was collected for analysis of this outcome measure.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Physician Assessment of Spasticity
Description: as for outcome 1
Time Frame: Month 12
Population: Planned analysis: All participants. Not enough data was collected for analysis of this outcome measure.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events were not collected/assessed for this study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Not enough data was collected for analysis of Physician's Assessment of Spasticity outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.